CLINICAL TRIAL: NCT05323188
Title: Evaluation of Basal Tryptasemia According to Age in a Pediatric Control Population
Brief Title: Serum Basal Tryptase Levels in Healthy Children
Acronym: KID-Tryp
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220353
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Basal Tryptasemia
Keywords: Serum basal tryptase levels; Pediatric control population; Basal tryptasemia according to age; Basal tryptasemia according to sex; Mastocytosis; Mast cell activation syndromes (MCAS)
MeSH Terms: conditions — Mastocytosis; Mast Cell Activation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 120µL of plasma to assay the tryptase; after the tryptase assay, the tube will be systematically discarded, there will be no biospecimens retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects: Control pediatric population: no excess of chronic inflammatory or allergic disease compared to the general French population.
  Interventions: Other: Tryptase dosage

INTERVENTIONS:
Other: Tryptase dosage — Collection of biological waste from a blood test for complete blood count (CBC) of care. Centrifugation to recover the plasma, then dosage of the tryptase.

SUMMARY:
The National REference Center for MASTocytosis (CEREMAST), located at the Necker-Enfants Malades Hospital, is particularly interested in two groups of rare diseases whose common point is excessive activation of mast cells: mastocytosis and mast cell activation syndromes (MCAS). Unlike MCAS, whose symptoms result solely from this aberrant mast cell activation, in mastocytosis there is, in addition, an expansion and a clonal accumulation of mast cells in different target organs. These two diseases are heterogeneous in their clinical presentation and can begin in early childhood. While the diagnostic criteria for mastocytosis are well established, those for MCAS are unclear, causing major diagnostic error and therefore poor patient care.

To date, there is no study evaluating tryptase standards in children less than 18 years of age.

The research focuses on the dosage of tryptase in a control population of children aged 0 to 18 years.

Each patient receiving a complete blood count (CBC) in a surgery department of the Necker-Enfants Malades hospital will be selected to participate in the study. After the CBC analysis, the rest of the sample will be kept for this research instead of being discarded.

Knowing the norms of tryptase according to age would be an important tool for dermatologists, allergists and pediatricians caring for patients suspected of MCAS or mastocytosis. A blood test could thus avoid a few years of diagnostic wandering in the MCAS and mastocytosis.

DETAILED DESCRIPTION:
The National REference Center for MASTocytosis (CEREMAST), located at the Necker-Enfants Malades Hospital, is particularly interested in two groups of rare diseases whose common point is excessive activation of mast cells: mastocytosis and mast cell activation syndromes (MCAS). Unlike MCAS, whose symptoms result solely from this aberrant mast cell activation, in mastocytosis there is, in addition, an expansion and a clonal accumulation of mast cells in different target organs. These two diseases are heterogeneous in their clinical presentation and can begin in early childhood. While the diagnostic criteria for mastocytosis are well established, those for MCAS are unclear, causing major diagnostic error and therefore poor patient care.

At CEREMAST, for the pediatric branch, just over 700 children with mastocytosis and 150 with MCAS are followed. For each patient, a tryptase assay is performed. Over the years, CEREMAST is able to confirm that the standard of tryptase currently given as <11.4µg/L is not valid in children and clearly objectify that the level of normal tryptase increases with age in the child. Several patients with MCAS with hereditary hyper-alpha-tryptasemia (HAT) are followed at CEREMAST with diagnostic delays of 4 years on average. The knowledge among the doctors who took care of these patients that a tryptase at 7µg/L can be pathological in children could have avoided this wandering, and allowed the faster implementation of an effective antihistamine treatment.

Recent studies have shown that familial hypertryptasemia or hereditary hyper-alpha-tryptasemia (HAT) of autosomal dominant transmission was associated with an increase in the number of copies of the TPSAB1 gene, coding for tryptase alpha 1 and beta. By now systematically looking for amplifications of the TPSAB1 gene in all CEREMAST patients, it has been noted that a duplication may be associated with a tryptase at 6 μg/L, considered normal in children.

To date, there is no study evaluating tryptase standards in children less than 18 years of age.

The research focuses on the dosage of tryptase in a control population of children aged 0 to 18 years.

Each patient receiving a complete blood count (CBC) in a surgery department of the Necker-Enfants Malades hospital will be selected to participate in the study. After the CBC analysis, the rest of the sample will be kept for this research instead of being discarded.

Knowing the norms of tryptase according to age would be an important tool for dermatologists, allergists and pediatricians caring for patients suspected of MCAS or mastocytosis. A blood test could thus avoid a few years of diagnostic wandering in the MCASs and mastocytosis.

ELIGIBILITY:
Inclusion Criteria:

* Minor patients aged 0-18
* Patient for whom a complete blood count (CBC) is carried out for their care in a surgery department (orthopedic, visceral, maxillofacial, neurology, cardiology surgery) at the Necker-Enfants Malades hospital
* Information and non-opposition of the subjects and of holders of parental authority subjects

Exclusion Criteria:

- Patients hospitalized in departments other than surgery at Necker-Enfants Malades Hospital

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients for whom a complete blood count (CBC) is carried out for their care in a surgery department (orthopedic, visceral, maxillofacial, neurology, cardiology surgery) at the Necker-Enfants Malades hospital, in order to have a control pediatric population with no excess of chronic inflammatory or allergic disease compared to the general French population.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Serum basal tryptase levels according to age | 8 months
  Basal tryptasemia according to age in a pediatric control population.

SECONDARY OUTCOMES:
Serum basal tryptasemia levels according to sex | 8 months
  Basal tryptasemia according to sex in a pediatric control population.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Polivka, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Luc de Chaisemartin, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puel M, Rossignol J, Devin C, Madrange M, Diep A, Roland PN, Chollet-Martin S, Husson J, Hermine O, Bodemer C, Brouzes C, De Chaisemartin L, Polivka L; CEREMAST network. Redefining tryptase norms in the pediatric population reveals sex-based differences: Clinical implications. Allergy. 2025 Jan;80(1):335-338. doi: 10.1111/all.16365. Epub 2024 Oct 19. No abstract available. PMID 39425617